CLINICAL TRIAL: NCT06026605
Title: A MulticenterOpen LableDose Escalat Tion and Dose Expansion Clinical Study to Evaluate the Safety, Tolerance and Ini Itial Effectiveness of WTX212A Injection in Patients with Unresectable or Metasta Atic Advanced Solid Tumors
Brief Title: A Dose Escalation and Dose Expansion Trial of WTX212A in the Treatment of Patients with Advanced Malignant Tumors
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Zhejiang University (Other)
Responsible Party: Principal Investigator, TingBo Liang, Professor, Zhejiang University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Reboot-102
Record Dates: First submitted 2023-08-21; First posted 2023-09-07 (Actual); Last update posted 2025-01-16 (Actual); Status verified 2024-05

CONDITIONS: Unresectable or Metastatic Advanced Solid Tumors

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- WTX212A (Experimental): WTX212A infusion once every 21 days
  Interventions: Drug: WTX212A

INTERVENTIONS:
Drug: WTX212A — WTX212A infusion once every 21 days

SUMMARY:
This trial is a multi-center, open-label investigator-initiated clinical study (IIT) to evaluate the safety, pharmacokinetics, pharmacodynamics and effectiveness of WTX212A injection in the treatment of patients with unresectable or metastatic advanced solid tumors who failed in previous systematic therapy.

The study was divided into two phases: dose escalation and dose expansion

DETAILED DESCRIPTION:
The study was divided into two phases: dose escalation and dose expansion Detailed Description: This trial is a multi-center, open-label investigator-initiated clinical study(llT)to evaluate the safety, pharmacokinetics, pharmacodynamics and effectiveness of WTX212A injection in the treatment of patients with unresectable or metastatic advanced solid tumors who failed in previous systematic therapy.

ELIGIBILITY:
Inclusion Criteria:

* 1. Must signs an informed consent form, understands this study, is willing to follow and has the ability to complete all experimental procedures; 2. Aged 18 to 75 years old (including threshold); 3. Histopathology diagnosed unresectable or metastatic solid tumors who have failed systemic treatment or have no effective standard treatment, or who are unwilling to accept standard treatment or are not suitable for standard treatment; 4. ECOG≤1； 5. Expected life ≥ 3 months； 6. Male participants, their spouses, and female participants of childbearing age should agree to use a medically recognized effective contraceptive method from the signing of the informed consent form until 3 months after the last administration; 7. Women of childbearing age must have a negative pregnancy testing results within ≤ 7 days before the first trial drug administration.

Exclusion Criteria:

- 1. Other serious medical diseases, including but not limited to: uncontrolled diabetes, active peptic ulcer, active bleeding, etc., and people with uncontrollable or serious cardiovascular diseases, 2. Pleural and ascitic fluids with clinical symptoms and the need for repeated drainage; 3. Previous or recent history of pulmonary fibrosis, severe lung function damage caused by pneumoconiosis, radiation pneumonia, and drug-related pneumonia; 4. History of adverse events related to the use of IO drugs that require permanent cessation of IO treatment; 5. Known to have other malignant tumors, currently progressing or completing treatment at least once in the past 3 years.

6. Symptomatic central nervous system (CNS) metastasis confirmed by imaging or pathological examination and clinically unstable for at least 14 days prior to enrollment who require steroid treatment; 7. Hereditary bleeding tendencies or coagulation disorders, or a history of thrombosis, hemolysis, or hemorrhagic diseases; 8. Received significant surgical treatment or obvious traumatic injury within 28 days prior to the start of research treatment;

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Estimated)
Dates: Start 2023-08-25 (Actual); Primary Completion 2026-08-30 (Estimated); Study Completion 2026-08-30 (Estimated)

PRIMARY OUTCOMES:
incidence of adverse events | through study completion, an average of 1 year
  The incidence of Adverse Events during the treatment of WTX212A injection
incidence of treatment related adverse events (TRAE) | through study completion, an average of 1 year
  The incidence of TRAE during the treatment of WTX212A injection
incidence of severe adverse events (SAE) | through study completion, an average of 1 year
  The incidence of SAE during the treatment of WTX212A injection

SECONDARY OUTCOMES:
Cmax | through study completion, an average of 1 months
  Cmax
Tmax | through study completion, an average of 1 months
  Tmax
AUC0-t | through study completion, an average of 1 months
  AUC0-t
t1/2 | through study completion, an average of 1 months
  t1/2
CL | through study completion, an average of 1 months
  CL
Cmin,ss | through study completion, an average of 1 months
  Cmin,ss
Cmax,ss | through study completion, an average of 1 months
  Cmax,ss
Tmax,ss | through study completion, an average of 1 months
  Tmax,ss
AUC（0-τ）ss. | through study completion, an average of 1 months
  AUC（0-τ）ss.
the occupancy rate of PD-1 receptor on the surface of peripheral blood T cells | through study completion, an average of 1 year
  the occupancy rate of PD-1 receptor on the surface of peripheral blood T cells in subjects after WTX212A infusion
Objecive Response Rate (ORR) | through study completion, an average of 4 months
  According to Response Evaluation Criteria In Solid Tumors Version 1.1
Anti-drug antibody (ADA) | through study completion, an average of 1 year
  escribe the number and percentage of anti-drug antibodies (ADA) produced by subjects at each time point after treatment, and the time of producing ADA

OTHER OUTCOMES:
Anti-drug antibodies (ADA) | through study completion, an average of 1 year
  The proportion of anti-drug antibodies (ADA) after WTX212A infusion
The absolute value of immune cell subsets | through study completion, an average of 1 year
  The absolute value of immune cell subsets
The percentage of immune cell subsets | through study completion, an average of 1 year
  The percentage of immune cell subsets
The proportion of PD-L1 expression in tumor cells/immune cells | through study completion, an average of 1 year
  The proportion of PD-L1 expression in tumor cells/immune cells

CONTACTS AND LOCATIONS:
Locations (1):
- the First Affiliated Hospital, School of Medicine, Zhejiang University, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No